CLINICAL TRIAL: NCT00234728
Title: An Open-Label, Bilaterally-Controlled Single Center Study to Compare the Efficacy of Occlusion of Topical Agents With a Hydrophilic Occlusive Dressing to Treatment With Occlusive Dressing Without the Addition of Topical Agents
Brief Title: Study of a New Dressing for Use With Topical Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teikoku Pharma USA, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPU-2005-02
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2008-07-02 (Estimated); Status verified 2008-06

CONDITIONS: Psoriasis
Keywords: psoriasis; hydrogel; occlusive dressing; occlusion; hydrocortisone; tacrolimus; Protopic; triamcinolone; calcipotriene; Dovonex; halobetasol; Ultravate
MeSH Terms: conditions — Psoriasis; Bites and Stings | interventions — Occlusive Dressings

INTERVENTIONS:
Device: Occlusive dressing

SUMMARY:
The purpose of this study is to determine if a new dressing designed to be used with topical medications will enhance the effects of these topical medications.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed the informed consent form and HIPAA authorization form
* Male or female subject at least 18 years of age
* A diagnosis of stable plaque-type psoriasis vulgaris with at least one "mirror image" pair of symmetric lesions on either the trunk, arms, or legs that would serve as target lesions. Paired target lesions must be in similar anatomic locations (e.g., right and left elbows or right and left knees) and have roughly equal (no more than one point difference) modified PASI scores. Both paired target lesions must have PASI scores equal to or greater than 1.5
* Any additional diagnoses must, in the investigator's opinion, not preclude the subject from safely participating in this study or interfere with the evaluation of the subject's psoriasis
* Psoriasis must be clinically stable for at least 30 days before enrollment
* Subject is able to completely discontinue the use of any medication or therapy for relief of psoriasis in the target areas to be treated
* Subject is able to completely discontinue the use of any systemic medication or therapy (e.g. oral or injectable psoriasis medications, PUVA phototherapy, herbal remedies, or acupuncture) for relief of psoriasis
* Female subjects must be postmenopausal (defined as one year without menses), physically incapable of becoming pregnant, or using an acceptable birth control method. Acceptable methods of birth control include hormonal contraceptives or double-barrier methods (condom, diaphragm with spermicidal agent or IUD). If practicing an acceptable method of birth control, the subject must have confirmation of a negative urine pregnancy test at Screening
* Subject must be reliable and mentally competent to complete study measurements
* Subject is able to understand and agrees to comply with study requirements, attend study visits, and comply with the restrictions during the study.

Exclusion Criteria:

* Subject has a skin disorder other than psoriasis in the target areas to be evaluated
* Known hypersensitivity to any component of the test medications
* Pigmentation, extensive scarring, or pigmented lesions in affected areas that would interfere with evaluation of efficacy parameters
* Clinically infected psoriasis at baseline
* Subject is pregnant or nursing
* Guttate, pustular, erythrodermic, or other non-plaque forms of psoriasis
* Spontaneously worsening or improving psoriasis within 30 days of enrollment
* Any evidence of atrophy in the areas selected for treatment with topical corticosteroid
* History of treating potential target lesions differently from one another
* Topical or intralesional therapies (other than emollients) or UVB phototherapy on potential target lesions within two weeks of starting study treatment
* Systemic therapy, PUVA phototherapy, or a systemic investigational therapy for psoriasis within 30 days prior to study entry
* Treatment with topical investigational therapy of the target lesions within 30 days prior to study entry
* Subject is considered unreliable as to medication compliance or adherence to scheduled appointments as determined by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-09; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of topical medications with new occlusive dressing at baseline, weeks 2, 4, 6, 8.

SECONDARY OUTCOMES:
Efficacy with new occlusive dressing alone without topical medications at baseline, weeks 2, 4, 6, 8.

CONTACTS AND LOCATIONS:
Overall Officials: John Koo, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Psoriasis and Skin Treatment Center, San Francisco, California, United States